CLINICAL TRIAL: NCT00333606
Title: Effects of Acupuncture on the Auditory Evoked Potentials: a Randomized Volunteer Crossover Study
Brief Title: Acupuncture and Auditory Evoked Potentials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taras Usichenko (Other)
Responsible Party: Sponsor-Investigator, Taras Usichenko, Dr. Taras Usichenko, University Medicine Greifswald
Organization: University Medicine Greifswald (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: III UV 12/06
Record Dates: First submitted 2006-06-03; First posted 2006-06-06 (Estimated); Results first posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2017-04

CONDITIONS: Evoked Potentials; Healthy Volunteers
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Verum acupuncture (Experimental): Acupuncture of specific acupuncture points
  Interventions: Behavioral: Acupuncture
- Sham acupuncture (Sham Comparator): Acupuncture of non-specific acupuncture points
  Interventions: Behavioral: Acupuncture

INTERVENTIONS:
Behavioral: Acupuncture — Body acupuncture of 1 specific point per trial session

SUMMARY:
To investigate whether body acupuncture of acupuncture points specific for hearing influences the auditory avoked potentials in comparison to puncture of non-specific acupuncture points

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers aged 20-40 years
2. Physical status I according to American Society of Anesthesiologists (ASA) classification
3. No history of nervous or psychiatric disease
4. Normal audiogram before the study
5. No chronic consume of analgesics, anticoagulants and/or antiplatelet agents, sedatives or alcohol
6. No local infection at the site of acupuncture
7. Volunteers who have given informed consent

Exclusion Criteria:

1. Pregnant or nursing females.
2. History of peripheral neuropathy
3. Abnormal skin conditions (infection, scars, psoriasis, eczema)
4. Inflamed site of acupuncture within 1 week

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2005-01; Primary Completion 2007-02 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taras I Usichenko, M.D., Study Chair — Ernst Moritz Arndt University; Reinhard Schmidt, M.D., Principal Investigator — Ernst Moritz Arndt University
Locations (1):
- Ernst Moritz Arndt University, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was the crossover study with 60 participants. Each participant underwent 2 conditions: verum and sham acupuncture within an interval of at least one week.
Groups:
- Sham, Then Verum Acupuncture: Stimulation was applied to sham acupuncture point
- Verum, Then Sham Acupuncture: Stimulation was applied to verum acupuncture point
Period: Overall Study
Arm/Group | Sham, Then Verum Acupuncture | Verum, Then Sham Acupuncture
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Healthy volunteers
Groups:
- Verum, Then Sham Acupuncture: verum acupuncture means stimulation of specific acupuncture points
- Sham, Then Verum Acupuncture: Sham acupuncture means stimulation of non-specific points
- Total: Total of all reporting groups
Arm/Group | Verum, Then Sham Acupuncture | Sham, Then Verum Acupuncture | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  Germany | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Latencies of Auditory Evoked Potentials
Time Frame: before acupuncture stimulation
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Verum Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 60 | 60
ms | 255 (55) | 255 (55)

2. Secondary Outcome: Pain Intensity
Description: Visual Analogue Scale 0-100 mm, where 0=no pain, and 100=maximal pain
Time Frame: 30 min
Measure: Median (Inter-Quartile Range); unit: mm
Groups:
- Sham Acupuncture: Sham acupuncture means stimulation of non-specific points
- Verum Acupuncture: Acupuncture needles applied to specific acupuncture points
Arm/Group | Sham Acupuncture | Verum Acupuncture
Number analyzed (Participants) | 60 | 60
mm | 40 [10 to 60] | 20 [10 to 30]

ADVERSE EVENTS:
Time Frame: 2 weeks
Groups:
- Verum Acupuncture: verum acupuncture means stimulation of specific acupuncture points
Arm/Group | Verum Acupuncture | Sham Acupuncture
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No